CLINICAL TRIAL: NCT00017589
Title: Phase II Study of Genasense (Bcl-2 Antisense) Combined With Mylotarg (Gemtuzumab Ozogamicin) in Elderly Patients With Relapsed Acute Myeloid Leukemia
Brief Title: Oblimersen and Gemtuzumab Ozogamicin in Treating Older Patients With Relapsed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genta Incorporated (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068721; GENTA-GA210; UCCRC-10928
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2003-04

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — oblimersen; Gemtuzumab

INTERVENTIONS:
Biological: oblimersen sodium
Drug: gemtuzumab ozogamicin

SUMMARY:
RATIONALE: Monoclonal antibodies such as gemtuzumab ozogamicin can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Oblimersen may help gemtuzumab ozogamicin kill more cancer cells by making cancer cells more sensitive to the drug.

PURPOSE: Phase II trial to study the effectiveness of combining oblimersen and gemtuzumab ozogamicin in treating older patients who have relapsed acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the complete response rate of elderly patients with relapsed CD33-positive acute myeloid leukemia treated with oblimersen and gemtuzumab ozogamicin.
* Determine the overall response rate and duration of response of patients treated with this regimen.
* Determine the safety of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive oblimersen IV continuously on days 1-7 and 15-22 and gemtuzumab ozogamicin IV over 2 hours on days 4 and 18.

Patients are followed monthly for 6 months.

PROJECTED ACCRUAL: A total of 20-100 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed CD33+ acute myeloid leukemia (AML)

  * In first relapse from chemotherapy
  * Complete response lasting at least 3 months before relapse
* No CNS leukemia
* No secondary leukemia or history of antecedent hematologic disorder prior to initial onset of AML (e.g., myelodysplasia)

PATIENT CHARACTERISTICS:

Age:

* 60 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC less than 30,000/mm^3
* No bleeding or coagulation disorder except disease-related disseminated intravascular coagulation

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* PT and PTT no greater than 1.5 times upper limit of normal OR
* INR no greater than 1.3
* No history of chronic hepatitis or cirrhosis

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No uncontrolled congestive heart failure
* No New York Heart Association class III or IV heart disease

Pulmonary:

* No severe pulmonary disease

Other:

* HIV negative
* No other concurrent medical disease that would preclude study entry
* No known hypersensitivity to phosphorothioate-containing oligonucleotides, gemtuzumab ozogamicin or any of its components, E. coli protein, or any product produced in E. coli
* No other concurrent malignancy
* No known human anti-human antibodies
* No uncontrolled seizure disorder
* No active uncontrolled infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior allogeneic or autologous stem cell transplantation
* No prior therapy with an anti-CD33 antibody (e.g., gemtuzumab ozogamicin or M195)

Chemotherapy:

* See Disease Characteristics
* At least 2 weeks since prior cancer chemotherapy except intrathecal chemotherapy or hydroxyurea

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 2 weeks since prior systemic radiotherapy

Surgery:

* At least 2 weeks since prior major surgery
* No prior organ allograft

Other:

* At least 3 weeks since prior antileukemic therapy and recovered
* No other concurrent investigational therapy
* No concurrent immunosuppressive therapy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-12; Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley R. Frankel, MD, Study Chair — Genta Incorporated
Locations (1):
- Genta Incorporated, Berkeley Heights, New Jersey, United States

REFERENCES:
- [Result] Moore J, Seiter K, Kolitz J, Stock W, Giles F, Kalaycio M, Zenk D, Marcucci G. A Phase II study of Bcl-2 antisense (oblimersen sodium) combined with gemtuzumab ozogamicin in older patients with acute myeloid leukemia in first relapse. Leuk Res. 2006 Jul;30(7):777-83. doi: 10.1016/j.leukres.2005.10.025. Epub 2006 May 26. PMID 16730060